CLINICAL TRIAL: NCT04470492
Title: Study on Prevention and Treatment of Atherosclerotic Cerebral Occlusive Disease With Remote Ischemic Conditioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, VP, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RICO
Record Dates: First submitted 2020-07-06; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Atherosclerosis
Keywords: cerebral atherosclerotic occlusion; remote ischemic conditioning; ischemic stroke
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental)
  Interventions: Combination Product: Doctormate®+Medical Management
- Control (Other)
  Interventions: Drug: Medical Management

INTERVENTIONS:
Combination Product: Doctormate®+Medical Management — Patients will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (200mmHg) twice daily and conventional medication for 3 months.
  Arms: Experiment
Drug: Medical Management — Patients will be treated with conventional medication for 3 months.
  Arms: Control

SUMMARY:
The primary objective of the study will be to determine whether remote limb ischemic conditioning (RLIC) together with conventional medication therapy compared with only medication therapy reduces the 3-month risk of composite cardio-cerebral vascular event in patients with a recent TIA or IS caused by occlusion of a cerebral artery.

After screening period, eligible patients will be randomly allocated into 2 groups.In addition, all participants receive an usual clinical therapy.

DETAILED DESCRIPTION:
In this study, Patients in the RLIC group will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (200mmHg) twice daily and conventional medication; patients in the control group will be treated only with conventional medication. In the study, the RLIC treatment will be comprised of 5 cycles of bilateral upper limb ischemia and reperfusion, which will be induced by 2 cuffs placed around the upper arms respectively and inflated to 200mmHg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age from 40 to 80 years old.
2. Patients with cerebral arterial occlusion which have been confirmed by CTA, MRA, or other evidence (including intracranial and extracranial arterial occlusion), and there is no indication of intervention and surgery, and at the same time the patients combined more than two risk factors for atherosclerosis.
3. The entry event is acute ischemic cerebrovascular disease (TIA or cerebral infarction), of which the condition was relatively stable within 30 days of onset, and mRS≤4.
4. Informed consent obtained.

Exclusion Criteria:

1. Thrombolytic therapy within 24 hours prior to enrollment.
2. Progressive neurological signs within 24 hours prior to enrollment.
3. Cerebral venous thrombosis/stenosis.
4. Intracranial arterial occlusion due to arterial dissection, Moya Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid (CSF) pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus.
5. Any of the following unequivocal cardiac source of embolism: rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with the participation.
6. Uncontrolled severe hypertension [sitting systolic blood pressure (SBP) >180 mmHg and/or sitting diastolic blood pressure (DBP) >110 mmHg after medication].
7. Patients with abnormal laboratory parameters: aspartate transaminase (AST) and/or alanine transaminase (ALT) >3×upper limit of normal range; creatinine clearance <0.6 ml/s and/or serum creatinine >265 μmol/l (>3.0 mg/dl); platelets <100×109/L.
8. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural) within 90 days prior to enrollment.
9. Intracranial neoplasm, cerebral aneurysm or arteriovenous malformation.
10. Known retinal hemorrhage or visceral bleeding within 30 days prior to enrollment.
11. Severe hemostatic disorder or severe coagulation dysfunction.
12. Subclavian arterial stenosis≥50% or subclavian steal syndrome.
13. Extracranial stenosis ≥50%.
14. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform one of these procedures within 12 months after enrollment.
15. Major surgery (including open femoral, aortic, or carotid surgery, cardiac) within previous 30 days or scheduled in the 12 months after enrollment.
16. Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
17. Life expectancy<3 years.
18. Pregnant or breast-feeding women.
19. Unwilling to be followed up or poor compliance for treatment.
20. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.
21. Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
3-month composite cardio-cerebral vascular event rate | During the first 3 months from randomization.

SECONDARY OUTCOMES:
Recurrence of TIA or infarction rate in the area of responsible vessel domination within 3 months | During the first 3 months from randomization.
Changes in National Institutes of Health Stroke Scale(NIHSS) within 3 months | During the first 3 months from randomization.
Changes in modified Rankin Scale(mRS) within 3 months | During the first 3 months from randomization.
Changes in Barthel Index(BI) within 3 months | During the first 3 months from randomization.
12-month composite cardio-cerebral vascular event rate | During the first 12 months from randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD.PhD, Principal Investigator — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided